CLINICAL TRIAL: NCT01005212
Title: Evaluation of Contrast-Enhanced Ultrasound to Detect Endoleaks After Endovascular Aortic Aneurysm Repair
Acronym: AAA CEUS
Status: Completed | Type: Observational
Sponsor: E. Peden, MD (Other)
Collaborators: Lantheus Medical Imaging (Industry); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, E. Peden, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00001211; 1007-0202 (Other: HMRI IRB)
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Endoleaks
Keywords: EVAR; Ultrasounds; AAA; endoleaks after endovascular repair of AAA
MeSH Terms: conditions — Endoleak | interventions — perflutren

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Definity — An intravenous line will be placed and 1.3 mL of the ultrasound contrast agent DEFINITY® will be added to 50 mL sterile saline. Flow will be initiated at 4.0 mL/minute and adjusted for optimal imaging. A maximum of 1.3 mL or one vial of ultrasound contrast will be used per patient per session according to the manufacturer's guidelines.

SUMMARY:
This study will be a cross-sectional survey of interobserver variability associated with contrast enhanced ultrasound (CEUS) to detect endoleaks using computed tomographic angiography (CTA) as the practice standard. The investigators will enroll 40 consecutive patients undergoing endovascular abdominal aortic aneurysm repair (EVAR). At the first follow-up visit after the procedure, participants will undergo two abdominal ultrasound examinations with and without contrast, and one CTA. Analyses will be conducted to examine interobserver variability in the detection and characterization of endoleaks using contrast-enhanced ultrasound (CEUS). Other endpoints include examination of sensitivity and specificity of CEUS compared to CTA, and characterization of the number and types of endoleaks detected.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or greater;
2. Diagnosed with abdominal aortic aneurysm and has undergone or is scheduled to undergo endovascular repair procedure.
3. Has not completed the first scheduled post-treatment follow-up exam
4. Voluntary participation and signature of IRB-approved informed consent.

Exclusion Criteria:

1. Inability to consent (includes non-English speaking patients)
2. Has already completed the first scheduled post-treatment follow-up exam.
3. Clinical instability;
4. Pregnancy / breast feeding;
5. Known allergy to perflutren;
6. Known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts (based on manufacturer recommendations for use);
7. Recent heart attack (<6 months), unstable angina or uncontrolled cardiopulmonary disease
8. Clinically unstable or recent worsening congestive heart failure (based on FDA warning)
9. Serious ventricular arrhythmias or at high risk for arrhythmias
10. Respiratory failure (based on FDA warning)
11. Severe emphysema, pulmonary emboli or other conditions that compromise pulmonary arterial vasculature (based on FDA warning)
12. Any reason judged by the investigators to hamper inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects that have undgone endovascular repair of abdominal aortic aneurysms (EVAR).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Peden, MD, Principal Investigator — Houston Methodist Hosptial
Locations (2):
- United States (2):
  - Houston Methodist Hospital; Department of Cardiovascualr Surgery, Houston, Texas
  - Houston Methodist Hospital; Department of Cardiovascular Surgery, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baum RA, Carpenter JP, Cope C, Golden MA, Velazquez OC, Neschis DG, Mitchell ME, Barker CF, Fairman RM. Aneurysm sac pressure measurements after endovascular repair of abdominal aortic aneurysms. J Vasc Surg. 2001 Jan;33(1):32-41. doi: 10.1067/mva.2001.111807. PMID 11137921
- [Background] Baum RA, Carpenter JP, Stavropoulous SW, Fairman RM. Diagnosis and management of type 2 endoleaks after endovascular aneurysm repair. Tech Vasc Interv Radiol. 2001 Dec;4(4):222-6. doi: 10.1016/s1089-2516(01)90012-5. PMID 11894049
- [Background] Bargellini I, Napoli V, Petruzzi P, Cioni R, Vignali C, Sardella SG, Ferrari M, Bartolozzi C. Type II lumbar endoleaks: hemodynamic differentiation by contrast-enhanced ultrasound scanning and influence on aneurysm enlargement after endovascular aneurysm repair. J Vasc Surg. 2005 Jan;41(1):10-8. doi: 10.1016/j.jvs.2004.10.037. PMID 15696037
- [Background] Bendick PJ, Bove PG, Long GW, Zelenock GB, Brown OW, Shanley CJ. Efficacy of ultrasound scan contrast agents in the noninvasive follow-up of aortic stent grafts. J Vasc Surg. 2003 Feb;37(2):381-5. doi: 10.1067/mva.2003.17. PMID 12563210
- [Background] Bromley PJ, Kaufman JA. Abdominal aortic aneurysms before and after endograft implantation: evaluation by computed tomography. Tech Vasc Interv Radiol. 2001 Mar;4(1):15-26. doi: 10.1053/tvir.2001.23090. PMID 11981786
- [Background] Carrafiello G, Recaldini C, Lagana D, Piffaretti G, Fugazzola C. Endoleak detection and classification after endovascular treatment of abdominal aortic aneurysm: value of CEUS over CTA. Abdom Imaging. 2008 May-Jun;33(3):357-62. doi: 10.1007/s00261-007-9268-3. PMID 17619925
- [Background] Chuter TA, Faruqi RM, Sawhney R, Reilly LM, Kerlan RB, Canto CJ, Lukaszewicz GC, Laberge JM, Wilson MW, Gordon RL, Wall SD, Rapp J, Messina LM. Endoleak after endovascular repair of abdominal aortic aneurysm. J Vasc Surg. 2001 Jul;34(1):98-105. doi: 10.1067/mva.2001.111487. PMID 11436081
- [Background] Dill-Macky MJ, Wilson SR, Sternbach Y, Kachura J, Lindsay T. Detecting endoleaks in aortic endografts using contrast-enhanced sonography. AJR Am J Roentgenol. 2007 Mar;188(3):W262-8. doi: 10.2214/AJR.05.0532. PMID 17312033
- [Background] Deaton DH, Makaroun MS, Fairman RM. Endoleak: predictive value for aneurysm growth at 3 years. Ann Vasc Surg. 2002 Jan;16(1):37-42. doi: 10.1007/s10016-001-0129-1. Epub 2002 Jan 16. PMID 11904802
- [Background] Eskandari MK, Yao JS, Pearce WH, Rutherford RB, Veith FJ, Harris P, Bernhard VM, Becker GJ, Morasch MD, Chrisman HB, Ryu RK, Matsumura JS. Surveillance after endoluminal repair of abdominal aortic aneurysms. Cardiovasc Surg. 2001 Oct;9(5):469-71. doi: 10.1016/s0967-2109(01)00044-8. No abstract available. PMID 11489651
- [Background] Giannoni MF, Palombo G, Sbarigia E, Speziale F, Zaccaria A, Fiorani P. Contrast-enhanced ultrasound imaging for aortic stent-graft surveillance. J Endovasc Ther. 2003 Apr;10(2):208-17. doi: 10.1177/152660280301000208. PMID 12877601
- [Background] Giannoni MF, Fanelli F, Citone M, Cristina Acconcia M, Speziale F, Gossetti B. Contrast ultrasound imaging: the best method to detect type II endoleak during endovascular aneurysm repair follow-up. Interact Cardiovasc Thorac Surg. 2007 Jun;6(3):359-62. doi: 10.1510/icvts.2006.137265. Epub 2007 Jan 8. PMID 17669866
- [Background] Henao EA, Hodge MD, Felkai DD, McCollum CH, Noon GP, Lin PH, Lumsden AB, Bush RL. Contrast-enhanced Duplex surveillance after endovascular abdominal aortic aneurysm repair: improved efficacy using a continuous infusion technique. J Vasc Surg. 2006 Feb;43(2):259-64; discussion 264. doi: 10.1016/j.jvs.2005.09.045. PMID 16476596
- [Background] Heilberger P, Schunn C, Ritter W, Weber S, Raithel D. Postoperative color flow duplex scanning in aortic endografting. J Endovasc Surg. 1997 Aug;4(3):262-71. doi: 10.1177/152660289700400305. PMID 9291051
- [Background] Hiatt MD, Rubin GD. Surveillance for endoleaks: how to detect all of them. Semin Vasc Surg. 2004 Dec;17(4):268-78. doi: 10.1053/j.semvascsurg.2004.09.003. PMID 15614750
- [Background] Jaakkola P, Hippelainen M, Farin P, Rytkonen H, Kainulainen S, Partanen K. Interobserver variability in measuring the dimensions of the abdominal aorta: comparison of ultrasound and computed tomography. Eur J Vasc Endovasc Surg. 1996 Aug;12(2):230-7. doi: 10.1016/s1078-5884(96)80112-2. PMID 8760988
- [Background] Jones WB, Taylor SM, Kalbaugh CA, Joels CS, Blackhurst DW, Langan EM 3rd, Gray BH, Youkey JR. Lost to follow-up: a potential under-appreciated limitation of endovascular aneurysm repair. J Vasc Surg. 2007 Sep;46(3):434-40; discussion 440-1. doi: 10.1016/j.jvs.2007.05.002. PMID 17826228
- [Background] McWilliams RG, Martin J, White D, Gould DA, Rowlands PC, Haycox A, Brennan J, Gilling-Smith GL, Harris PL. Detection of endoleak with enhanced ultrasound imaging: comparison with biphasic computed tomography. J Endovasc Ther. 2002 Apr;9(2):170-9. doi: 10.1177/152660280200900206. PMID 12010096
- [Background] Muthu C, Gordon M, Buckenham T, Lewis D. The case for lifelong follow-up after endovascular aneurysm repair. N Z Med J. 2005 Nov 11;118(1225):U1729. No abstract available. PMID 16286942
- [Background] Napoli V, Bargellini I, Sardella SG, Petruzzi P, Cioni R, Vignali C, Ferrari M, Bartolozzi C. Abdominal aortic aneurysm: contrast-enhanced US for missed endoleaks after endoluminal repair. Radiology. 2004 Oct;233(1):217-25. doi: 10.1148/radiol.2331031767. PMID 15454621
- [Background] Resch T, Ivancev K, Brunkwall J, Nyman U, Malina M, Lindblad B. Distal migration of stent-grafts after endovascular repair of abdominal aortic aneurysms. J Vasc Interv Radiol. 1999 Mar;10(3):257-64; discussion 265-6. doi: 10.1016/s1051-0443(99)70027-8. PMID 10102188
- [Background] Rydberg J, Lalka S, Johnson M, Cikrit D, Dalsing M, Sawchuk A, Shafique S. Characterization of endoleaks by dynamic computed tomographic angiography. Am J Surg. 2004 Nov;188(5):538-43. doi: 10.1016/j.amjsurg.2004.07.011. PMID 15546566
- [Background] Sawhney R, Kerlan RK, Wall SD, Chuter TA, Ruiz DE, Canto CJ, LaBerge JM, Reilly LM, Yee J, Wilson MW, Jean-Claude J, Faruqi RM, Gordon RL. Analysis of initial CT findings after endovascular repair of abdominal aortic aneurysm. Radiology. 2001 Jul;220(1):157-60. doi: 10.1148/radiology.220.1.r01jl22157. PMID 11425989
- [Background] Singh K, Jacobsen BK, Solberg S, Bonaa KH, Kumar S, Bajic R, Arnesen E. Intra- and interobserver variability in the measurements of abdominal aortic and common iliac artery diameter with computed tomography. The Tromso study. Eur J Vasc Endovasc Surg. 2003 May;25(5):399-407. doi: 10.1053/ejvs.2002.1856. PMID 12713777
- [Background] Singh K, Jacobsen BK, Solberg S, Kumar S, Arnesen E. The difference between ultrasound and computed tomography (CT) measurements of aortic diameter increases with aortic diameter: analysis of axial images of abdominal aortic and common iliac artery diameter in normal and aneurysmal aortas. The Tromso Study, 1994-1995. Eur J Vasc Endovasc Surg. 2004 Aug;28(2):158-67. doi: 10.1016/j.ejvs.2004.03.018. PMID 15234697
- [Background] Tillich M, Hausegger KA, Tiesenhausen K, Tauss J, Groell R, Szolar DH. Helical CT angiography of stent-grafts in abdominal aortic aneurysms: morphologic changes and complications. Radiographics. 1999 Nov-Dec;19(6):1573-83. doi: 10.1148/radiographics.19.6.g99no091573. PMID 10555675
- [Background] Wanhainen A, Bergqvist D, Bjorck M. Measuring the abdominal aorta with ultrasonography and computed tomography - difference and variability. Eur J Vasc Endovasc Surg. 2002 Nov;24(5):428-34. doi: 10.1053/ejvs.2002.1748. PMID 12435343
- [Background] White GH, Yu W, May J, Chaufour X, Stephen MS. Endoleak as a complication of endoluminal grafting of abdominal aortic aneurysms: classification, incidence, diagnosis, and management. J Endovasc Surg. 1997 May;4(2):152-68. doi: 10.1177/152660289700400207. PMID 9185003
- [Background] White GH, May J, Petrasek P, Waugh R, Stephen M, Harris J. Endotension: an explanation for continued AAA growth after successful endoluminal repair. J Endovasc Surg. 1999 Nov;6(4):308-15. doi: 10.1583/1074-6218(1999)0062.0.CO;2. PMID 10893130

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: study recruitment ended
Period: Overall Study
Arm/Group | Single Arm
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: AAA patients
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 70 [50 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Endoleak Detection
Description: Persistent of a pulsatile intrasac color flow outside the stent-graft
Time Frame: Same day outcome
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm: Patients undergoig post-EVAR follow-up with CEUS
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Participants | 9

ADVERSE EVENTS:
Groups:
- CEUS-Single Arm: Patients undergoing post-EVAR surveillance with CEUS
Arm/Group | CEUS-Single Arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No